CLINICAL TRIAL: NCT01329757
Title: Efficacy and Safety of Growth Hormone (GH) Treatment in Spinal Cord Injury(SCI): A Triple-blinded, Randomised, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Growth Hormone Treatment in Spinal Cord Injury
Acronym: GHSCI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Nacional de Parapléjicos de Toledo (Other)
Collaborators: Ministerio de Salud y Politicas Sociales (Ministry of Health) (Unknown)
Responsible Party: Principal Investigator, Antonio Oliviero, MD, PhD, Neurologist, Hospital Nacional de Parapléjicos de Toledo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FHNP-CT001
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Growth Hormone; Trauma; Incomplete; ASIA
MeSH Terms: conditions — Spinal Cord Injuries; Wounds and Injuries | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GH (Active Comparator): Administration of a daily dose of GH (0.4mg)for 1 year
  Interventions: Drug: GH
- Placebo (Placebo Comparator): Administration of a daily dose of placebo for 1 year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GH — Administration of a subcutaneously injected daily dose of GH (0.4mg)for 1 year
  Other Names: Genotonorm
  Arms: GH
Drug: Placebo — Administration of a subcutaneously injected daily dose of placebo for 1 year
  Other Names: Provided by the Genotonorm producer (Pfizer)
  Arms: Placebo

SUMMARY:
Objectives: To evaluate the efficacy and safety of one year treatment based on daily doses of exogenous growth hormone (GH) in patients with traumatic spinal cord injury. The first six months the pharmacological treatment will be associated to rehabilitation treatment.

The main hypothesis is that GH can improve motor function of patients with traumatic spinal cord injury below the lesion level. The hypothesis is based on possible effects of GH at muscle and synaptic level. GH can also promote axonal growth and regeneration.

Design: Clinical trial placebo-controlled, double-blind intervention with blind evaluation by third parties and blinding in the analysis of data (triple-blind design).

Duration of intervention and monitoring: 364 days.

Primary outcome measures. Changes of the American Spinal Injury Association (ASIA) scale (motor score)

ELIGIBILITY:
Inclusion Criteria:

* Traumatic Spinal cord injury
* Incomplete (ASIA scale B or C)
* Level of injury: Between C4 and D12
* More than 18 months from the SCI injury.

Exclusion Criteria:

* Non traumatic Spinal cord injury
* Complete SCI (ASIA A)
* Incomplete (ASIA D or E)
* Less than 18 months from the SCI
* Intensive Care Unit (ICU) staying for a period of 2 months or more
* More than 3 urological infections in the last year
* Pneumonia in the 6 months prior to the study
* Severe respiratory failure
* History of head trauma
* Severe psychiatric disorder
* A history of heart disease, diabetes or hypertension
* Concomitant Neurological Diseases
* Regular use of substances of abuse
* Patients with severe kidney and / or liver failure.
* Patients who can not be included in an intensive rehabilitation program
* Patients who are pregnant or breast-feeding
* History of malignancy
* Impossibility to obtain informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Motor Score of the American Spinal Injury Association (ASIA) scale | 12 months
  Motor score of the ASIA scale reports the strenght of 10 key muscles in each body side (5 key muscles in upper limb and 5 key muscles in lower limb). The strenght is rated between 0 and 5 (Medical Research Council-MRC scale). The ASIA motor score range is between 0 and 100 (normal).

SECONDARY OUTCOMES:
ASIA | 12 months
  ASIA grades
ASIA sensory score | 12 months
  ASIA sensory score
Spasticity | Baseline, 15 days, 6 months, 12 months
  Penn scale and Ashworth scale
Pain | Baseline, 15 days, 6 months, 12 months
  Visual analogic scale (VAS)
Independence Measures and Quality of life | 12 months
  Spinal Cord Indipendence Measures (SCIM) and the Quality of Life Questionnaire (EQ 5D)
Neurophysiological Measures | 6 months and 12 months
  Motor Evoked Potentials, Somatosensory Evoked Potentials, Motor Neurography
Safety | 15, 30, 60, 90, 120, 150, 180, 360 days
  Recording of any adverse event, full blood and urine examination

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Oliviero, MD, PhD, Principal Investigator — Hospital Nacional de Paraplejicos
Locations (1):
- Hospital Nacional de Paraplejicos, Toledo, Spain